CLINICAL TRIAL: NCT01386684
Title: Canadian Real-Life Evaluation of the Effectiveness of Lupron in the Management of Prostate Cancer (CRONOS)
Brief Title: Real Life Evaluation of Lupron in the Management of Prostate Cancer: A Canadian Post Marketing Observational Study
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: JSS Medical Research Inc. (Industry); CMX Research (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-811
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Prostate Cancer: Patients with prostate cancer who were receiving treatment with leuprolide acetate (Lupron).

SUMMARY:
The purpose of this study is to evaluate the Canadian Real Life Evaluation of the Effectiveness of Lupron in the Management of Prostate Cancer.

DETAILED DESCRIPTION:
This is a Canadian Post Marketing Observational Study utilizing a prospective cohort design. Patients with Prostate Cancer who are prescribed Lupron will be entered into the study cohort and will be followed for a maximum of 36 months with recommended assessments at 3, 6, 12, 18, 24, 30 and 36 months after baseline. Treatment of the patients and follow up will be according to the physician's judgment, regional regulations and the product monograph.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent allowing the use of their data for the study and providing permission for contact by the study personnel
* Diagnosed with Prostate Cancer
* Prescribed Lupron as part of his treatment by his treating physician

Exclusion Criteria:

* Currently participating in another prospective study including controlled clinical trials and observational studies.
* Patient cannot or will not sign informed consent
* Survival expectancy less than 2-3 years as per the treating physician's judgment
* Presence of other condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of Prostate Cancer
* History of alcohol or drug abuse
* No longer than 6 months of therapy if currently on luteinizing hormone-releasing hormone (LHRH) treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from the offices of university or community urologists/oncologists across Canada treating patients with PCa.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Pelizon, MD, Study Director — AbbVie Corporation

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Prostate Cancer: Patients with prostate cancer who were receiving treatment with Lupron.
Period: Overall Study
Arm/Group | Patients With Prostate Cancer
Started | 552
Completed | 259
Not Completed | 293
Not completed — Lost to Follow-up | 51
Not completed — Other | 51
Not completed — Death | 47
Not completed — Withdrawal of Consent | 44
Not completed — Alternative Therapy Required | 37
Not completed — Disease Progression | 28
Not completed — Adverse Event | 20
Not completed — Noncompliance | 8
Not completed — Protocol Violation | 4
Not completed — Missing | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 552

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Defined as the Time From Patient Recruitment to Biochemical Progression Based on Doubling of Prostate Specific Antigen (PSA) Velocity or PSA > 5.0
Description: PFS defined as the time from patient recruitment to biochemical progression based on doubling of prostate specific antigen (PSA) velocity or PSA > 5.0, objective tumor progression (RECIST criteria), or death. The distribution of PFS was estimated using Kaplan-Meier methodology. The point estimate and standard error (SE) of the distribution are provided.
Time Frame: 36 months
Measure: Mean (Standard Error); unit: months
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
months | 20.76 (0.59)

2. Primary Outcome: Progression-free Survival (PFS) Defined as the Time From Patient Recruitment to a Change to an Absolute Value of PSA > 2 ng/mL on at Least 2 Consecutive Tests
Description: A second definition of PFS was used due to changes in the definition of biochemical progression: the time from patient recruitment to a change to an absolute value of PSA > 2 ng/mL on at least 2 consecutive tests, objective tumor progression (RECIST criteria), or death. The distribution of PFS was estimated using Kaplan-Meier methodology. The point estimate and standard error (SE) of the distribution are provided.
Time Frame: 36 months
Measure: Mean (Standard Error); unit: months
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
months | 21.89 (0.69)

3. Secondary Outcome: Castration Resistant Prostate Cancer (CRPC): Number of Participants
Description: CRPC defined as PSA > 2 ng/mL on at least 2 consecutive tests.
Time Frame: 36 months
Population: All participants who achieved PSA levels ≤ 2 ng/mL
Measure: Number; unit: participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 440
participants | 84

4. Secondary Outcome: Castration Resistant Prostate Cancer (CRPC): Time to Event
Description: CRPC defined as PSA > 2 ng/mL on at least 2 consecutive tests. The distribution of time to CRPC was estimated using Kaplan-Meier methodology. The point estimate and standard error of the distribution are provided.
Time Frame: 36 months
Population: All participants who achieved PSA levels ≤2 ng/mL
Measure: Mean (Standard Error); unit: months
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 440
months | 26.01 (0.42)

5. Secondary Outcome: Total Serum Testosterone: Percentage of Participants With ≤ 0.7 Nmol/L, > 0.7 to ≤ 1.7 Nmol/L, and > 1.7 Nmol/L at Each Visit
Description: Total serum testosterone was assessed at each study visit. The percentage of participants with total serum testosterone ≤ 0.7 nmol/L, > 0.7 to ≤ 1.7 nmol/L, and > 1.7 nmol/L are provided at each time point.
Time Frame: Months 0 (Baseline), 3, 6, 12, 18, 24, 30, and 36
Population: All participants with available data at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
percentage of participants
  Month 0: ≤ 0.7 nmol/L: number analyzed (Participants) | 190
  Month 0: ≤ 0.7 nmol/L | 16.3
  Month 3: ≤ 0.7 nmol/L: number analyzed (Participants) | 245
  Month 3: ≤ 0.7 nmol/L | 65.3
  Month 6: ≤ 0.7 nmol/L: number analyzed (Participants) | 229
  Month 6: ≤ 0.7 nmol/L | 62.9
  Month 12: ≤ 0.7 nmol/L: number analyzed (Participants) | 208
  Month 12: ≤ 0.7 nmol/L | 68.8
  Month 18: ≤ 0.7 nmol/L: number analyzed (Participants) | 187
  Month 18: ≤ 0.7 nmol/L | 69.0
  Month 24: ≤ 0.7 nmol/L: number analyzed (Participants) | 160
  Month 24: ≤ 0.7 nmol/L | 68.8
  Month 30: ≤ 0.7 nmol/L: number analyzed (Participants) | 133
  Month 30: ≤ 0.7 nmol/L | 69.2
  Month 36: ≤ 0.7 nmol/L: number analyzed (Participants) | 122
  Month 36: ≤ 0.7 nmol/L | 55.7
  Month 0: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 190
  Month 0: > 0.7 to ≤ 1.7 nmol/L | 6.3
  Month 3: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 245
  Month 3: > 0.7 to ≤ 1.7 nmol/L | 32.7
  Month 6: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 229
  Month 6: > 0.7 to ≤ 1.7 nmol/L | 31.4
  Month 12: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 208
  Month 12: > 0.7 to ≤ 1.7 nmol/L | 18.8
  Month 18: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 187
  Month 18: > 0.7 to ≤ 1.7 nmol/L | 15.5
  Month 24: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 160
  Month 24: > 0.7 to ≤ 1.7 nmol/L | 12.5
  Month 30: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 133
  Month 30: > 0.7 to ≤ 1.7 nmol/L | 12.8
  Month 36: > 0.7 to ≤ 1.7 nmol/L: number analyzed (Participants) | 122
  Month 36: > 0.7 to ≤ 1.7 nmol/L | 15.6
  Month 0: > 1.7 nmol/L: number analyzed (Participants) | 190
  Month 0: > 1.7 nmol/L | 77.4
  Month 3: > 1.7 nmol/L: number analyzed (Participants) | 245
  Month 3: > 1.7 nmol/L | 2.0
  Month 6: > 1.7 nmol/L: number analyzed (Participants) | 229
  Month 6: > 1.7 nmol/L | 5.7
  Month 12: > 1.7 nmol/L: number analyzed (Participants) | 208
  Month 12: > 1.7 nmol/L | 12.5
  Month 18: > 1.7 nmol/L: number analyzed (Participants) | 187
  Month 18: > 1.7 nmol/L | 15.5
  Month 24: > 1.7 nmol/L: number analyzed (Participants) | 160
  Month 24: > 1.7 nmol/L | 18.8
  Month 30: > 1.7 nmol/L: number analyzed (Participants) | 133
  Month 30: > 1.7 nmol/L | 18.0
  Month 36: > 1.7 nmol/L: number analyzed (Participants) | 122
  Month 36: > 1.7 nmol/L | 28.7

6. Secondary Outcome: Total Serum Testosterone Levels at Each Visit
Description: Total serum testosterone was assessed at each study visit.
Time Frame: Months 0 (Baseline), 3, 6, 12, 18, 24, 30, and 36
Population: All participants with available data at given time point.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
nmol/L
  Month 0: number analyzed (Participants) | 190
  Month 0 | 10.9 (8.90)
  Month 3: number analyzed (Participants) | 245
  Month 3 | 0.6 (0.98)
  Month 6: number analyzed (Participants) | 229
  Month 6 | 1.0 (2.32)
  Month 12: number analyzed (Participants) | 208
  Month 12 | 1.5 (3.29)
  Month 18: number analyzed (Participants) | 187
  Month 18 | 1.9 (4.05)
  Month 24: number analyzed (Participants) | 160
  Month 24 | 2.1 (4.31)
  Month 30: number analyzed (Participants) | 133
  Month 30 | 2.3 (4.81)
  Month 36: number analyzed (Participants) | 122
  Month 36 | 2.9 (4.69)

7. Secondary Outcome: Total Serum Testosterone: Time to Increase Over Castrate Levels
Description: Total serum testosterone was assessed at each study visit. The time to increased total serum testosterone over the castrate levels (>1.7 nmol/L) are provided. The distribution of time to increase in total serum testosterone levels was estimated using Kaplan-Meier methodology. The point estimate and standard error (SE) of the distribution are provided.
Time Frame: 36 months
Population: All participants who achieved castrate testosterone levels (≤1.7 nmol/L)
Measure: Mean (Standard Error); unit: months
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 359
months | 31.20 (0.67)

8. Secondary Outcome: Prostatic Specific Antigen (PSA): Percentage of Participants With Serum PSA < 1 ng/mL, 1 to < 5 ng/mL, 5 to < 10 ng/mL, and ≥10 ng/mL at Each Visit
Description: Serum PSA was assessed at each study visit. The percentage of participants with serum PSA < 1 ng/mL, 1 to < 5 ng/mL, 5 to < 10 ng/mL, and ≥10 ng/mL are provided at each time point.
Time Frame: Months 0 (Baseline), 3, 6, 12, 18, 24, 30, and 36
Population: All participants with available date at given time point
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
percentage of participants
  Month 0: <1 ng/mL: number analyzed (Participants) | 545
  Month 0: <1 ng/mL | 15.2
  Month 3: <1 ng/mL: number analyzed (Participants) | 440
  Month 3: <1 ng/mL | 55.9
  Month 6: <1 ng/mL: number analyzed (Participants) | 432
  Month 6: <1 ng/mL | 61.8
  Month 12: <1 ng/mL: number analyzed (Participants) | 387
  Month 12: <1 ng/mL | 63.6
  Month 18: <1 ng/mL: number analyzed (Participants) | 336
  Month 18: <1 ng/mL | 64.6
  Month 24: <1 ng/mL: number analyzed (Participants) | 280
  Month 24: <1 ng/mL | 60.7
  Month 30: <1 ng/mL: number analyzed (Participants) | 253
  Month 30: <1 ng/mL | 56.9
  Month 36: <1 ng/mL: number analyzed (Participants) | 233
  Month 36: <1 ng/mL | 57.5
  Month 0: 1 to <5 ng/mL: number analyzed (Participants) | 545
  Month 0: 1 to <5 ng/mL | 17.4
  Month 3: 1 to <5 ng/mL: number analyzed (Participants) | 440
  Month 3: 1 to <5 ng/mL | 31.4
  Month 6: 1 to <5 ng/mL: number analyzed (Participants) | 432
  Month 6: 1 to <5 ng/mL | 21.5
  Month 12: 1 to <5 ng/mL: number analyzed (Participants) | 387
  Month 12: 1 to <5 ng/mL | 16.8
  Month 18: 1 to <5 ng/mL: number analyzed (Participants) | 336
  Month 18: 1 to <5 ng/mL | 17.9
  Month 24: 1 to <5 ng/mL: number analyzed (Participants) | 280
  Month 24: 1 to <5 ng/mL | 16.4
  Month 30: 1 to <5 ng/mL: number analyzed (Participants) | 253
  Month 30: 1 to <5 ng/mL | 19.8
  Month 36: 1 to <5 ng/mL: number analyzed (Participants) | 233
  Month 36: 1 to <5 ng/mL | 18.9
  Month 0: 5 to <10 ng/mL: number analyzed (Participants) | 545
  Month 0: 5 to <10 ng/mL | 17.6
  Month 3: 5 to <10 ng/mL: number analyzed (Participants) | 440
  Month 3: 5 to <10 ng/mL | 4.1
  Month 6: 5 to <10 ng/mL: number analyzed (Participants) | 432
  Month 6: 5 to <10 ng/mL | 7.6
  Month 12: 5 to <10 ng/mL: number analyzed (Participants) | 387
  Month 12: 5 to <10 ng/mL | 7.5
  Month 18: 5 to <10 ng/mL: number analyzed (Participants) | 336
  Month 18: 5 to <10 ng/mL | 8.9
  Month 24: 5 to <10 ng/mL: number analyzed (Participants) | 280
  Month 24: 5 to <10 ng/mL | 6.8
  Month 30: 5 to <10 ng/mL: number analyzed (Participants) | 253
  Month 30: 5 to <10 ng/mL | 7.5
  Month 36: 5 to <10 ng/mL: number analyzed (Participants) | 233
  Month 36: 5 to <10 ng/mL | 9.0
  Month 0: ≥10 ng/mL: number analyzed (Participants) | 545
  Month 0: ≥10 ng/mL | 49.7
  Month 3: ≥10 ng/mL: number analyzed (Participants) | 440
  Month 3: ≥10 ng/mL | 8.6
  Month 6: ≥10 ng/mL: number analyzed (Participants) | 432
  Month 6: ≥10 ng/mL | 9.0
  Month 12: ≥10 ng/mL: number analyzed (Participants) | 387
  Month 12: ≥10 ng/mL | 12.1
  Month 18: ≥10 ng/mL: number analyzed (Participants) | 336
  Month 18: ≥10 ng/mL | 8.6
  Month 24: ≥10 ng/mL: number analyzed (Participants) | 280
  Month 24: ≥10 ng/mL | 16.1
  Month 30: ≥10 ng/mL: number analyzed (Participants) | 253
  Month 30: ≥10 ng/mL | 15.8
  Month 36: ≥10 ng/mL: number analyzed (Participants) | 233
  Month 36: ≥10 ng/mL | 14.6

9. Secondary Outcome: Prostatic Specific Antigen (PSA) Levels at Each Visit
Description: Serum PSA was assessed at each study visit.
Time Frame: Months 0 (Baseline), 3, 6, 12, 18, 24, 30, and 36
Population: All participants with available data at given time point.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
ng/ml
  Month 0: number analyzed (Participants) | 545
  Month 0 | 65.0 (377.60)
  Month 3: number analyzed (Participants) | 440
  Month 3 | 6.5 (41.33)
  Month 6: number analyzed (Participants) | 432
  Month 6 | 12.0 (80.64)
  Month 12: number analyzed (Participants) | 387
  Month 12 | 19.1 (128.51)
  Month 18: number analyzed (Participants) | 336
  Month 18 | 13.3 (113.98)
  Month 24: number analyzed (Participants) | 280
  Month 24 | 11.2 (56.69)
  Month 30: number analyzed (Participants) | 253
  Month 30 | 13.5 (65.79)
  Month 36: number analyzed (Participants) | 233
  Month 36 | 8.2 (37.12)

10. Secondary Outcome: Functional Assessment of Cancer Therapy Questionnaire - General (FACT-G) Total Score: Change From Baseline to Each Visit
Description: The FACT-G questionnaire is used with patients of any tumor type to assess patient quality of life (QoL). FACT-G is a self-administered, 28-item questionnaire assessing physical, functional, social and emotional well-being, as well as patient satisfaction with treatment. All questions in the FACT-G use a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much). The FACT-G total score is computed as the sum of the four subscale scores and has a possible range of 0-108. Higher scores indicate better QoL. Change in FACT-G was analyzed using repeated measures mixed effects general linear model (GLM). A positive change from baseline indicates improved QoL.
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
units on a scale
  Month 3 | -0.9 (0.6)
  Month 6 | -2.2 (0.6)
  Month 12 | -1.7 (0.6)
  Month 18 | -1.0 (0.7)
  Month 24 | -1.4 (0.7)
  Month 30 | -1.3 (0.7)
  Month 36 | -1.9 (0.8)

11. Secondary Outcome: Functional Assessment of Cancer Therapy Questionnaire - Prostate Cancer (FACT-P) Total Score: Change From Baseline to Each Visit
Description: The FACT-P questionnaire is used with patients with prostate cancer to assess patient quality of life (QoL). FACT-P is a self-administered, 28-item questionnaire assessing physical, functional, social and emotional well-being, as well as patient satisfaction with treatment. All questions in the FACT-P use a 5-point rating scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; and 4 = very much). The FACT-P total score is computed as the sum of the four subscale scores and has a possible range of 0-108. Higher scores indicate better QoL. Change in FACT-P was analyzed using repeated measures mixed effects general linear model (GLM). A negative change from baseline indicates decreased QoL.
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
units on a scale
  Month 3 | -1.1 (0.8)
  Month 6 | -2.8 (0.8)
  Month 12 | -2.4 (0.9)
  Month 18 | -1.8 (0.9)
  Month 24 | -2.1 (0.9)
  Month 30 | -2.3 (1.0)
  Month 36 | -3.0 (1.0)

12. Secondary Outcome: International Index of Erectile Function (IIEF-5) Total Score: Change From Baseline to Each Visit
Description: IIEF-5 is a 5-item, self-administered questionnaire assessing the presence and severity of erectile dysfunction. A score of 1 (very low) to 5 (very high) is awarded to each of the 5 questions. The IIEF-5 total score is a sum of the responses to the 5 items. Total scores range from 5 to 25, with higher scores indicating less dysfunction. Change in IIEF-5 was analyzed using repeated measures mixed effects general linear model (GLM). A negative change from baseline indicates an increase in dysfunction.
Time Frame: Month 0 (Baseline) and Months 6, 12, 18, 24, 30, and 36
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
units on a scale
  Month 6 | -2.7 (0.3)
  Month 12 | -3.2 (0.3)
  Month 18 | -3.3 (0.3)
  Month 24 | -3.7 (0.3)
  Month 30 | -3.5 (0.3)
  Month 36 | -3.3 (0.3)

13. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants With Medical Insurance for Prescription Medications
Description: The Health Care Utilization and Health Economics Questionnaire is a descriptive, self-administered series of questions aimed at measuring the patient's health care utilization and economic impact of the disease. The questionnaire was used to assess since the last visit the frequency of physician visits; utilization of other health care professionals; visits to clinics, emergency rooms, and hospitalizations related to prostate cancer; use of prescription and non-prescription medications for the management of prostate cancer were determined; and out of pocket expenses for medications and health care.
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with available data at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 452
  Month 3 | 408
  Month 6 | 384
  Month 12 | 328
  Month 18 | 279
  Month 24 | 258
  Month 30 | 220
  Month 36 | 196

14. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Visited a Physician for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 38
  Month 3 | 44
  Month 6 | 38
  Month 12 | 34
  Month 18 | 20
  Month 24 | 23
  Month 30 | 14
  Month 36 | 8

15. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Visits With a Physician for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who had visited a physician and with available data at given time point.
Measure: Mean (Standard Deviation); unit: physician visits
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
physician visits
  Month 0: number analyzed (Participants) | 15
  Month 0 | 1.2 (0.56)
  Month 3: number analyzed (Participants) | 19
  Month 3 | 1.5 (0.84)
  Month 6: number analyzed (Participants) | 19
  Month 6 | 7.1 (13.93)
  Month 12: number analyzed (Participants) | 17
  Month 12 | 1.6 (1.17)
  Month 18: number analyzed (Participants) | 6
  Month 18 | 2.7 (1.86)
  Month 24: number analyzed (Participants) | 5
  Month 24 | 2.4 (1.14)
  Month 30: number analyzed (Participants) | 3
  Month 30 | 2.0 (1.00)
  Month 36: number analyzed (Participants) | 3
  Month 36 | 2.0 (0.00)

16. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Visited a Healthcare Professional for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 20
  Month 3 | 23
  Month 6 | 20
  Month 12 | 21
  Month 18 | 8
  Month 24 | 11
  Month 30 | 9
  Month 36 | 3

17. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Visits With a Healthcare Professional for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who had visited a healthcare professional and with available data at given time point.
Measure: Mean (Standard Deviation); unit: healthcare professional visits
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
healthcare professional visits
  Month 0: number analyzed (Participants) | 11
  Month 0 | 7.8 (14.05)
  Month 3: number analyzed (Participants) | 11
  Month 3 | 3.5 (4.11)
  Month 6: number analyzed (Participants) | 11
  Month 6 | 18.5 (19.06)
  Month 12: number analyzed (Participants) | 11
  Month 12 | 3.1 (2.12)
  Month 18: number analyzed (Participants) | 4
  Month 18 | 2.3 (0.96)
  Month 24: number analyzed (Participants) | 3
  Month 24 | 1.7 (1.15)
  Month 30: number analyzed (Participants) | 5
  Month 30 | 1.6 (0.89)
  Month 36: number analyzed (Participants) | 0

18. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Visited a Hospital Emergency Room for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 9
  Month 3 | 7
  Month 6 | 3
  Month 12 | 8
  Month 18 | 5
  Month 24 | 6
  Month 30 | 4
  Month 36 | 2

19. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Visits to A Hospital Emergency Room for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who had visited a hospital emergency room and with available data at given time point.
Measure: Mean (Standard Deviation); unit: hospital emergency room visits
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
hospital emergency room visits
  Month 0: number analyzed (Participants) | 5
  Month 0 | 1.2 (0.45)
  Month 3: number analyzed (Participants) | 1
  Month 3 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 6: number analyzed (Participants) | 1
  Month 6 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 12: number analyzed (Participants) | 5
  Month 12 | 1.4 (0.55)
  Month 18: number analyzed (Participants) | 1
  Month 18 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 24: number analyzed (Participants) | 0
  Month 30: number analyzed (Participants) | 2
  Month 30 | 1.0 (0.00)
  Month 36: number analyzed (Participants) | 0

20. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Used an Ambulance Service for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 4
  Month 3 | 2
  Month 6 | 4
  Month 12 | 2
  Month 18 | 2
  Month 24 | 3
  Month 30 | 2
  Month 36 | 1

21. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Times That an Ambulance Service Was Used for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who had used an ambulance service and with available data at given time point.
Measure: Mean (Standard Deviation); unit: ambulance service uses
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
ambulance service uses
  Month 0: number analyzed (Participants) | 1
  Month 0 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 3: number analyzed (Participants) | 0
  Month 6: number analyzed (Participants) | 1
  Month 6 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 12: number analyzed (Participants) | 0
  Month 18: number analyzed (Participants) | 1
  Month 18 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 24: number analyzed (Participants) | 0
  Month 30: number analyzed (Participants) | 1
  Month 30 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 36: number analyzed (Participants) | 0

22. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Visited Complementary/Alternate Therapy for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 3
  Month 3 | 2
  Month 6 | 1
  Month 12 | 4
  Month 18 | 3
  Month 24 | 0
  Month 30 | 0
  Month 36 | 1

23. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Visits For Complementary/Alternate Therapy for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who had visited complementary/alternate therapy and with available data at given time point.
Measure: Mean (Standard Deviation); unit: complementary/alternate therapy visits
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
complementary/alternate therapy visits
  Month 0: number analyzed (Participants) | 1
  Month 0 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 3: number analyzed (Participants) | 1
  Month 3 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 6: number analyzed (Participants) | 0
  Month 12: number analyzed (Participants) | 2
  Month 12 | 3.5 (2.12)
  Month 18: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0
  Month 30: number analyzed (Participants) | 0
  Month 36: number analyzed (Participants) | 0

24. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Used Any Other Medical Service for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 9
  Month 3 | 8
  Month 6 | 12
  Month 12 | 9
  Month 18 | 5
  Month 24 | 6
  Month 30 | 2
  Month 36 | 2

25. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Visits For Any Other Medical Service for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who had visited for any other medical service and with available data at given time point.
Measure: Mean (Standard Deviation); unit: visits for any other medical service
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
visits for any other medical service
  Month 0: number analyzed (Participants) | 5
  Month 0 | 7.4 (12.66)
  Month 3: number analyzed (Participants) | 4
  Month 3 | 2.0 (2.00)
  Month 6: number analyzed (Participants) | 1
  Month 6 | 1.0 (NA) — The estimated standard deviation of one sample is undefined
  Month 12: number analyzed (Participants) | 2
  Month 12 | 1.0 (0.00)
  Month 18: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0
  Month 30: number analyzed (Participants) | 0
  Month 36: number analyzed (Participants) | 1
  Month 36 | 1.0 (NA) — The estimated standard deviation of one sample is undefined

26. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Participants Who Were Admitted to the Hospital for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
Participants
  Month 0 | 29
  Month 3 | 14
  Month 6 | 9
  Month 12 | 14
  Month 18 | 9
  Month 24 | 5
  Month 30 | 4
  Month 36 | 8

27. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Number of Admissions to the Hospital for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants who were admitted to the hospital and with available data at given time point.
Measure: Mean (Standard Deviation); unit: admissions to the hospital
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
admissions to the hospital
  Month 0: number analyzed (Participants) | 29
  Month 0 | 1.0 (0.00)
  Month 3: number analyzed (Participants) | 14
  Month 3 | 1.0 (0.00)
  Month 6: number analyzed (Participants) | 9
  Month 6 | 1.0 (0.00)
  Month 12: number analyzed (Participants) | 14
  Month 12 | 1.0 (0.00)
  Month 18: number analyzed (Participants) | 9
  Month 18 | 1.0 (0.00)
  Month 24: number analyzed (Participants) | 5
  Month 24 | 1.0 (0.00)
  Month 30: number analyzed (Participants) | 4
  Month 30 | 1.0 (0.00)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 1.0 (0.00)

28. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Over-the-counter Medications for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for over-the-counter medications and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 368
  Month 0 | 21.5 (73.50)
  Month 3: number analyzed (Participants) | 327
  Month 3 | 19.3 (101.66)
  Month 6: number analyzed (Participants) | 298
  Month 6 | 25.5 (130.41)
  Month 12: number analyzed (Participants) | 254
  Month 12 | 26.6 (101.28)
  Month 18: number analyzed (Participants) | 223
  Month 18 | 20.9 (80.53)
  Month 24: number analyzed (Participants) | 197
  Month 24 | 13.9 (60.01)
  Month 30: number analyzed (Participants) | 167
  Month 30 | 13.4 (54.69)
  Month 36: number analyzed (Participants) | 152
  Month 36 | 13.1 (55.12)

29. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Payments to Health Care Professionals for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for payments to health care professionals and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 330
  Month 0 | 0.9 (11.66)
  Month 3: number analyzed (Participants) | 305
  Month 3 | 2.5 (30.24)
  Month 6: number analyzed (Participants) | 275
  Month 6 | 2.5 (31.18)
  Month 12: number analyzed (Participants) | 244
  Month 12 | 0.8 (12.80)
  Month 18: number analyzed (Participants) | 208
  Month 18 | 2.4 (34.67)
  Month 24: number analyzed (Participants) | 190
  Month 24 | 2.6 (36.27)
  Month 30: number analyzed (Participants) | 157
  Month 30 | 1.6 (19.95)
  Month 36: number analyzed (Participants) | 149
  Month 36 | 7.9 (62.50)

30. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Medical Procedures for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for medical procedures and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 337
  Month 0 | 14.0 (91.76)
  Month 3: number analyzed (Participants) | 304
  Month 3 | 2.6 (22.01)
  Month 6: number analyzed (Participants) | 278
  Month 6 | 4.1 (33.59)
  Month 12: number analyzed (Participants) | 246
  Month 12 | 3.0 (20.96)
  Month 18: number analyzed (Participants) | 211
  Month 18 | 2.7 (18.39)
  Month 24: number analyzed (Participants) | 189
  Month 24 | 6.8 (54.35)
  Month 30: number analyzed (Participants) | 158
  Month 30 | 5.2 (35.89)
  Month 36: number analyzed (Participants) | 149
  Month 36 | 2.9 (20.11)

31. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Payments for Medical Procedures or Laboratory Tests for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for payments for medical procedures or laboratory tests and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 337
  Month 0 | 14.0 (91.76)
  Month 3: number analyzed (Participants) | 304
  Month 3 | 2.6 (22.01)
  Month 6: number analyzed (Participants) | 278
  Month 6 | 4.1 (33.59)
  Month 12: number analyzed (Participants) | 246
  Month 12 | 3.0 (20.96)
  Month 18: number analyzed (Participants) | 211
  Month 18 | 2.7 (18.39)
  Month 24: number analyzed (Participants) | 189
  Month 24 | 6.8 (54.35)
  Month 30: number analyzed (Participants) | 158
  Month 30 | 5.2 (35.89)
  Month 36: number analyzed (Participants) | 149
  Month 36 | 2.9 (20.11)

32. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Medical Devices for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for medical devices and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 333
  Month 0 | 4.0 (40.46)
  Month 3: number analyzed (Participants) | 307
  Month 3 | 7.5 (58.00)
  Month 6: number analyzed (Participants) | 274
  Month 6 | 21.0 (292.53)
  Month 12: number analyzed (Participants) | 245
  Month 12 | 7.3 (96.50)
  Month 18: number analyzed (Participants) | 210
  Month 18 | 2.1 (16.79)
  Month 24: number analyzed (Participants) | 193
  Month 24 | 2.4 (22.88)
  Month 30: number analyzed (Participants) | 158
  Month 30 | 1.5 (12.96)
  Month 36: number analyzed (Participants) | 148
  Month 36 | 2.0 (24.66)

33. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Health Care or Extra Help At Home for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for health care or extra help at home and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 332
  Month 0 | 4.9 (58.06)
  Month 3: number analyzed (Participants) | 305
  Month 3 | 4.9 (60.31)
  Month 6: number analyzed (Participants) | 273
  Month 6 | 14.7 (189.44)
  Month 12: number analyzed (Participants) | 242
  Month 12 | 28.9 (390.75)
  Month 18: number analyzed (Participants) | 210
  Month 18 | 0.4 (6.21)
  Month 24: number analyzed (Participants) | 190
  Month 24 | 1.4 (14.26)
  Month 30: number analyzed (Participants) | 157
  Month 30 | 3.0 (24.16)
  Month 36: number analyzed (Participants) | 148
  Month 36 | 11.8 (92.40)

34. Secondary Outcome: Health Care Utilization and Health Economics Questionnaire: Out of Pocket Expenses for Transportation Costs for Prostate Cancer
Description: as for outcome 13
Time Frame: Month 0 (Baseline) and Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with out of pocket expenses for transportation costs and with available data at given time point.
Measure: Mean (Standard Deviation); unit: dollars (CAD)
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
dollars (CAD)
  Month 0: number analyzed (Participants) | 336
  Month 0 | 20.0 (124.86)
  Month 3: number analyzed (Participants) | 312
  Month 3 | 19.5 (77.92)
  Month 6: number analyzed (Participants) | 278
  Month 6 | 23.0 (96.03)
  Month 12: number analyzed (Participants) | 249
  Month 12 | 9.2 (27.87)
  Month 18: number analyzed (Participants) | 214
  Month 18 | 6.3 (19.88)
  Month 24: number analyzed (Participants) | 194
  Month 24 | 10.6 (87.22)
  Month 30: number analyzed (Participants) | 163
  Month 30 | 8.2 (26.54)
  Month 36: number analyzed (Participants) | 149
  Month 36 | 2.7 (9.30)

35. Secondary Outcome: Treatment Compliance
Description: Treatment compliance by participants was assessed as the number of missed injections since the last visit.
Time Frame: Months 3, 6, 12, 18, 24, 30, and 36
Population: All participants with available data at given time point.
Measure: Mean (Standard Deviation); unit: missed injections
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 552
missed injections
  Month 3: number analyzed (Participants) | 519
  Month 3 | 0.0 (0.12)
  Month 6: number analyzed (Participants) | 486
  Month 6 | 0.0 (0.17)
  Month 12: number analyzed (Participants) | 425
  Month 12 | 0.1 (0.35)
  Month 18: number analyzed (Participants) | 364
  Month 18 | 0.2 (0.53)
  Month 24: number analyzed (Participants) | 315
  Month 24 | 0.2 (0.66)
  Month 30: number analyzed (Participants) | 285
  Month 30 | 0.2 (0.57)
  Month 36: number analyzed (Participants) | 258
  Month 36 | 0.2 (0.83)

36. Secondary Outcome: Percentage of Participants With Changes in Current Prostate Cancer Treatment Since Last Visit.
Description: Participants were asked "Have there been any changes in the current prostate cancer treatment (not including Lupron) since last visit?"; if Yes, was the change "Initiation of new mediation/Change in Dose/Frequency" or "Discontinuation of medication". The percentage of subjects at each visit with a change in current prostate cancer treatment (Initiation or Change in Dose/Frequency or Discontinuation of Medication) is presented.
Time Frame: Months 3, 6, 12, 18, 24, 30, and 36
Population: The number of participants with changes in current prostate cancer treatment since the last visit at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Prostate Cancer
Number analyzed (Participants) | 522
percentage of participants
  Month 3 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 117
  Month 3 Initiation or Change in Dose/Frequency | 9.4
  Month 3 Discontinuation of Medication: number analyzed (Participants) | 117
  Month 3 Discontinuation of Medication | 90.6
  Month 6 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 47
  Month 6 Initiation or Change in Dose/Frequency | 42.6
  Month 6 Discontinuation of Medication: number analyzed (Participants) | 47
  Month 6 Discontinuation of Medication | 57.4
  Month 12 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 37
  Month 12 Initiation or Change in Dose/Frequency | 54.1
  Month 12 Discontinuation of Medication | 45.9
  Month 18 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 20
  Month 18 Initiation or Change in Dose/Frequency | 45.0
  Month 18 Discontinuation of Medication: number analyzed (Participants) | 20
  Month 18 Discontinuation of Medication | 45.0
  Month 24 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 25
  Month 24 Initiation or Change in Dose/Frequency | 60.0
  Month 24 Discontinuation of Medication: number analyzed (Participants) | 25
  Month 24 Discontinuation of Medication | 40.0
  Month 30 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 21
  Month 30 Initiation or Change in Dose/Frequency | 71.4
  Month 30 Discontinuation of Medication: number analyzed (Participants) | 21
  Month 30 Discontinuation of Medication | 28.6
  Month 36 Initiation or Change in Dose/Frequency: number analyzed (Participants) | 14
  Month 36 Initiation or Change in Dose/Frequency | 57.1
  Month 36 Discontinuation of Medication: number analyzed (Participants) | 14
  Month 36 Discontinuation of Medication | 42.9

ADVERSE EVENTS:
Time Frame: Spontaneously-reported adverse events (AEs) and serious adverse events (SAEs) were collected from the time that informed consent was given until 30 days following the last dose of physician-prescribed treatment (up to 37 months).
Arm/Group | Patients With Prostate Cancer
Serious Adverse Events (participants affected / at risk) | 132/552
Other Adverse Events (participants affected / at risk) | 77/552
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Prostate Cancer (N=552)
ANAEMIA (Blood and lymphatic system disorders) | 5
BANDAEMIA (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 4
ANGINA PECTORIS (Cardiac disorders) | 1
ANGINA UNSTABLE (Cardiac disorders) | 1
AORTIC VALVE STENOSIS (Cardiac disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 8
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 2
CARDIAC ARREST (Cardiac disorders) | 2
CARDIAC DISORDER (Cardiac disorders) | 2
CARDIAC FAILURE (Cardiac disorders) | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 9
CARDIOMEGALY (Cardiac disorders) | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 3
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 8
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2
PALPITATIONS (Cardiac disorders) | 1
SINUS BRADYCARDIA (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 3
DEAFNESS (Ear and labyrinth disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
DIPLOPIA (Eye disorders) | 1
OCULAR MYASTHENIA (Eye disorders) | 1
ABDOMINAL MASS (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 6
COELIAC DISEASE (Gastrointestinal disorders) | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1
DIVERTICULUM (Gastrointestinal disorders) | 1
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3
HAEMATEMESIS (Gastrointestinal disorders) | 1
HIATUS HERNIA (Gastrointestinal disorders) | 1
INTESTINAL MASS (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
ASTHENIA (General disorders) | 7
CHEST PAIN (General disorders) | 3
CHILLS (General disorders) | 1
CONDITION AGGRAVATED (General disorders) | 1
DEATH (General disorders) | 7
DISEASE PROGRESSION (General disorders) | 7
DRUG INEFFECTIVE (General disorders) | 1
FATIGUE (General disorders) | 4
GAIT DISTURBANCE (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4
IMPAIRED SELF-CARE (General disorders) | 1
INFLAMMATION (General disorders) | 1
LOCAL SWELLING (General disorders) | 1
MALAISE (General disorders) | 2
NO THERAPEUTIC RESPONSE (General disorders) | 1
OBSTRUCTION (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 2
PAIN (General disorders) | 4
PELVIC MASS (General disorders) | 1
PYREXIA (General disorders) | 5
UNEVALUABLE EVENT (General disorders) | 1
HEPATIC LESION (Hepatobiliary disorders) | 1
IMMUNOSUPPRESSION (Immune system disorders) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1
ESCHERICHIA INFECTION (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
GASTROENTERITIS ESCHERICHIA COLI (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 5
PYELONEPHRITIS ACUTE (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 3
SEPTIC SHOCK (Infections and infestations) | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 3
UROSEPSIS (Infections and infestations) | 3
ANAESTHETIC COMPLICATION (Injury, poisoning and procedural complications) | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2
FALL (Injury, poisoning and procedural complications) | 11
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 4
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1
TRACHEOSTOMY MALFUNCTION (Injury, poisoning and procedural complications) | 1
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1
BLOOD ALBUMIN DECREASED (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 2
BLOOD URINE PRESENT (Investigations) | 1
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 1
EJECTION FRACTION ABNORMAL (Investigations) | 1
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 2
EXERCISE ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
OXYGEN SATURATION DECREASED (Investigations) | 2
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1
SCAN MYOCARDIAL PERFUSION ABNORMAL (Investigations) | 2
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 1
TROPONIN INCREASED (Investigations) | 1
VENOUS PRESSURE JUGULAR INCREASED (Investigations) | 1
WEIGHT DECREASED (Investigations) | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
ACIDOSIS (Metabolism and nutrition disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
BILIARY NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HIGH GRADE B-CELL LYMPHOMA BURKITT-LIKE LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HORMONE-REFRACTORY PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
LUNG ADENOCARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO RECTUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14
PROSTATE CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA OF PHARYNX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BALANCE DISORDER (Nervous system disorders) | 2
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2
COMA (Nervous system disorders) | 1
DEMENTIA (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 3
HEADACHE (Nervous system disorders) | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 2
SEIZURE (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 4
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1
DEVICE OCCLUSION (Product Issues) | 1
ANXIETY (Psychiatric disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 3
DELIRIUM (Psychiatric disorders) | 3
DELUSION (Psychiatric disorders) | 1
DISORIENTATION (Psychiatric disorders) | 1
PARANOIA (Psychiatric disorders) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 6
CALCULUS BLADDER (Renal and urinary disorders) | 2
DYSURIA (Renal and urinary disorders) | 4
HAEMATURIA (Renal and urinary disorders) | 4
INCONTINENCE (Renal and urinary disorders) | 1
INTERCAPILLARY GLOMERULOSCLEROSIS (Renal and urinary disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 2
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 1
POLLAKIURIA (Renal and urinary disorders) | 1
RENAL CYST (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 4
URETERIC OBSTRUCTION (Renal and urinary disorders) | 1
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 3
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1
PROSTATOMEGALY (Reproductive system and breast disorders) | 1
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 3
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1
ACTIVITIES OF DAILY LIVING IMPAIRED (Social circumstances) | 1
BLADDER CALCULUS REMOVAL (Surgical and medical procedures) | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1
HYDROCELE OPERATION (Surgical and medical procedures) | 1
STERNOTOMY (Surgical and medical procedures) | 1
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 2
URINARY CYSTECTOMY (Surgical and medical procedures) | 1
ANGIOPATHY (Vascular disorders) | 1
AORTIC STENOSIS (Vascular disorders) | 1
BLEEDING VARICOSE VEIN (Vascular disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 4
HYPERTENSION (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Prostate Cancer (N=552)
LEUKOCYTE VACUOLISATION (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
EAR PAIN (Ear and labyrinth disorders) | 1
OCULAR MYASTHENIA (Eye disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 2
DYSPHAGIA (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 3
CHEST DISCOMFORT (General disorders) | 1
CHEST PAIN (General disorders) | 1
CHILLS (General disorders) | 2
DISEASE PROGRESSION (General disorders) | 1
DRUG INEFFECTIVE (General disorders) | 6
FATIGUE (General disorders) | 9
GAIT DISTURBANCE (General disorders) | 2
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3
INJECTION SITE ERYTHEMA (General disorders) | 1
INJECTION SITE PAIN (General disorders) | 1
INJECTION SITE REACTION (General disorders) | 1
INJECTION SITE SWELLING (General disorders) | 1
INJECTION SITE ULCER (General disorders) | 1
MALAISE (General disorders) | 1
NODULE (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
PAIN (General disorders) | 2
HEPATIC LESION (Hepatobiliary disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
DYSENTERY (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 2
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
RADIATION ASSOCIATED PAIN (Injury, poisoning and procedural complications) | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1
BLOOD CREATININE ABNORMAL (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 1
BLOOD TESTOSTERONE (Investigations) | 1
BLOOD TESTOSTERONE INCREASED (Investigations) | 1
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 1
HAEMOGLOBIN ABNORMAL (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 1
NEUTROPHIL TOXIC GRANULATION PRESENT (Investigations) | 1
OXYGEN SATURATION DECREASED (Investigations) | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 4
WEIGHT DECREASED (Investigations) | 1
WEIGHT INCREASED (Investigations) | 1
WHITE BLOOD CELL COUNT ABNORMAL (Investigations) | 1
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
CACHEXIA (Metabolism and nutrition disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1
FLUID INTAKE REDUCED (Metabolism and nutrition disorders) | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
HYPOPHAGIA (Metabolism and nutrition disorders) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
BONE LESION (Musculoskeletal and connective tissue disorders) | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1
JOINT DESTRUCTION (Musculoskeletal and connective tissue disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
WEIGHT BEARING DIFFICULTY (Musculoskeletal and connective tissue disorders) | 1
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
DEMENTIA (Nervous system disorders) | 2
DIZZINESS (Nervous system disorders) | 2
DYSGEUSIA (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 1
LETHARGY (Nervous system disorders) | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 1
NEURALGIA (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
TREMOR (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 2
DEPRESSION (Psychiatric disorders) | 1
EMOTIONAL DISORDER (Psychiatric disorders) | 1
EUPHORIC MOOD (Psychiatric disorders) | 1
LISTLESS (Psychiatric disorders) | 1
PSYCHIATRIC DECOMPENSATION (Psychiatric disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 2
NOCTURIA (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
PELVIC PAIN (Reproductive system and breast disorders) | 1
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RALES (Respiratory, thoracic and mediastinal disorders) | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1
ACTIVITIES OF DAILY LIVING IMPAIRED (Social circumstances) | 2
RADIOTHERAPY TO PROSTATE (Surgical and medical procedures) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 15
HYPOTENSION (Vascular disorders) | 2
PALLOR (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This was a real-world evidence assessment with clear limitations. One of the key limitations of the study was that treatment patterns were not fully documented. Furthermore, compliance/adherence may have impacted efficacy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.